CLINICAL TRIAL: NCT00000991
Title: A Randomized Trial of Three Anti-Pneumocystis Agents Plus Zidovudine for the Primary Prevention of Serious Infections in Patients With Advanced HIV Infection
Brief Title: A Study of Three Drugs Plus Zidovudine in the Prevention of Infections in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 081; 11056 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Toxoplasmosis; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Dapsone; Drug Evaluation; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine; Sulfamethoxazole-Trimethoprim
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Toxoplasmosis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Pentamidine; Trimethoprim, Sulfamethoxazole Drug Combination; Dapsone; Zidovudine

INTERVENTIONS:
Drug: Pentamidine isethionate
Drug: Sulfamethoxazole-Trimethoprim
Drug: Dapsone
Drug: Zidovudine

SUMMARY:
To evaluate and compare 3 anti-pneumocystis regimens plus zidovudine (AZT) in persons with HIV infection and T4 cell count less than 200 cells/mm3. All persons completing at least 8 weeks of therapy on 081 will be offered the opportunity to participate in the nested study (ACTG 981) of systemic antifungal therapy (fluconazole) versus local therapy (Clotrimazole) for the prevention of serious fungal disease.

Persons with HIV disease who are receiving AZT are at risk for PCP, toxoplasmosis, bacterial pneumonia, and other serious infections. It is therefore important to find drugs that can be given along with AZT to control these infections. Aerosolized pentamidine (PEN) has been shown to be useful in preventing PCP and is expected to lower the 2-year risk of PCP. Both sulfamethoxazole/trimethoprim (SMX/TMP) and dapsone probably also provide effective preventive treatment against PCP, and both may be useful in preventing toxoplasmosis and extrapulmonary pneumocystosis.

DETAILED DESCRIPTION:
Persons with HIV disease who are receiving AZT are at risk for PCP, toxoplasmosis, bacterial pneumonia, and other serious infections. It is therefore important to find drugs that can be given along with AZT to control these infections. Aerosolized pentamidine (PEN) has been shown to be useful in preventing PCP and is expected to lower the 2-year risk of PCP. Both sulfamethoxazole/trimethoprim (SMX/TMP) and dapsone probably also provide effective preventive treatment against PCP, and both may be useful in preventing toxoplasmosis and extrapulmonary pneumocystosis.

All patients receive AZT. In addition, they are placed in one of three groups to receive either SMX/TMP, dapsone, or PEN. Stratification criteria are:

Received first AZT equal to or less than 6 weeks prior to study entry. Received first AZT more than 6 weeks prior to study entry. Potential to participate in ACTG 981. ACTG center in which the patient is enrolled.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antifolate medication required to treat an intercurrent infection.
* Treatment of intercurrent infections or malignancies.
* Fluconazole.
* Itraconazole.
* Standard or investigational therapy for pneumocystosis (PCP) or toxoplasmosis.
* Only the forms of primary prophylaxis for PCP or toxoplasmosis assigned to the participant under the protocol. Patients who develop intolerance to all forms of prophylaxis assigned in this protocol or who develop PCP or toxoplasmosis may receive alternate or investigation forms of prophylaxis with or without zidovudine but must continue to be followed under this protocol.
* Discouraged but allowed: AL-721.
* Chronic acyclovir.
* Ketoconazole.
* Amphotericin B.
* Corticosteroids at greater than physiologic replacement doses are strongly discouraged.
* They should be used as briefly as possible and only for definite specific indications.

Patient must conform to the following:

* Receiving or candidates for zidovudine therapy at least 500 mg/day under current labeled indications with no history of pneumocystosis (PCP) or toxoplasmosis.
* Evidence of HIV infection documented by HIV antibody tests.
* T4 cell count less than 200 cells/mm3 at any time prior to study entry.
* Willing to sign informed consent.
* Willing to be followed by a participating ACTG center for duration of the study.
* Allowed: Concurrent enrollment in long-term follow-up studies in previously blinded trials of AZT (ACTG 016 and 019).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

* History of documented or presumed pneumocystosis (PCP) or toxoplasmosis.
* Active bacterial or mycobacterial infection.
* History of type I hypersensitivity, exfoliative rash, or rash with mucosal involvement, severe bronchospasm, or other life-threatening reaction to any of the study drugs or to other sulfas, sulfones, or pentamidine.
* History of intolerance causing dose interruption while receiving zidovudine at equal to or less than 600 mg/day or causing dose reduction to less than 500 mg/day within 4 weeks prior to entry.
* Advanced Kaposi's sarcoma or other malignancy not specifically allowed that has been rapidly progressive during the month prior to enrollment or which may be expected to require chemotherapy within 90 days of study entry.

Concurrent Medication:

Excluded:

* Active primary treatment for an infection or malignancy.
* Other form of antifolate medication not specifically allowed.
* Other antiretroviral or biologic response modifier.
* Ganciclovir, if it causes intolerance to AZT equal to or more than 500 mg/day.
* Foscarnet.

Patients with the following are excluded:

* Symptoms and conditions defined in Exclusion Coexisting Conditions.
* Glucose 6-phosphate dehydrogenase deficiency (GPD).
* History of pneumocystosis (PCP) or toxoplasmosis.
* History of type I hypersensitivity, exfoliative rash, or rash with mucosal involvement, severe bronchospasm, or other life-threatening reaction to any of the study drugs or to other sulfas, sulfones, or pentamidine.
* History of intolerance causing dose interruption while receiving zidovudine at equal to or less than 500 mg/day with 4 weeks pior to study entry.

Prior Medication:

Excluded within 4 weeks of study entry:

* Any other form of pneumocystosis (PCP) chemoprophylaxis.
* Active substance abuse, including alcohol.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Study Completion 1994-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S Bozzette, Study Chair; S Spector, Study Chair
Locations (21):
- United States (20):
  - USC CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - Ucsd, Avrc Crs, San Diego, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Chicago Children's CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Bozzette SA, Hays RD, Berry SH, Kanouse DE. A Perceived Health Index for use in persons with advanced HIV disease: derivation, reliability, and validity. Med Care. 1994 Jul;32(7):716-31. doi: 10.1097/00005650-199407000-00005. PMID 8028406
- [Background] Bozzette SA, Finkelstein DM, Spector SA, Frame P, Powderly WG, He W, Phillips L, Craven D, van der Horst C, Feinberg J. A randomized trial of three antipneumocystis agents in patients with advanced human immunodeficiency virus infection. NIAID AIDS Clinical Trials Group. N Engl J Med. 1995 Mar 16;332(11):693-9. doi: 10.1056/NEJM199503163321101. PMID 7854375
- [Background] Glick ME. CTG studies yield results. AIDS Clinical Trials Group. NIAID AIDS Agenda. 1995 Spring:8-9. PMID 11362451
- [Background] Justice AC, Rabeneck L, Hays RD, Wu AW, Bozzette SA. Sensitivity, specificity, reliability, and clinical validity of provider-reported symptoms: a comparison with self-reported symptoms. Outcomes Committee of the AIDS Clinical Trials Group. J Acquir Immune Defic Syndr. 1999 Jun 1;21(2):126-33. PMID 10360804
- [Background] Justice AC, Holmes W, Gifford AL, Rabeneck L, Zackin R, Sinclair G, Weissman S, Neidig J, Marcus C, Chesney M, Cohn SE, Wu AW; Adult AIDS Clinical Trials Unit Outcomes Committee. Development and validation of a self-completed HIV symptom index. J Clin Epidemiol. 2001 Dec;54 Suppl 1:S77-90. doi: 10.1016/s0895-4356(01)00449-8. PMID 11750213
- [Background] Ioannidis JP, Dixon DO, McIntosh M, Albert JM, Bozzette SA, Schnittman SM. Relationship between event rates and treatment effects in clinical site differences within multicenter trials: an example from primary Pneumocystis carinii prophylaxis. Control Clin Trials. 1999 Jun;20(3):253-66. doi: 10.1016/s0197-2456(98)00053-1. PMID 10357498
- [Background] DiRienzo AG, van Der Horst C, Finkelstein DM, Frame P, Bozzette SA, Tashima KT. Efficacy of trimethoprim-sulfamethoxazole for the prevention of bacterial infections in a randomized prophylaxis trial of patients with advanced HIV infection. AIDS Res Hum Retroviruses. 2002 Jan 20;18(2):89-94. doi: 10.1089/08892220252779629. PMID 11839141